CLINICAL TRIAL: NCT02409303
Title: A Screen-Refer-Treat (SRT) Model to Promote Earlier Access to ASD Intervention
Brief Title: An SRT Model for Early Access to ASD Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Wendy Stone, Professor of Psychology, University of Washington
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 47892; R01MH104302-01 (NIH)
Record Dates: First submitted 2015-03-26; First posted 2015-04-06 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Screening; Preventive intervention; Risk
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screen-Refer-Treat Intervention (Experimental): PCPs and EI Providers receive training workshops on validated, evidence-based practices (i.e., Online M-CHAT-R/F, STAT, and RIT) and then receive TA (i.e., Screen-Refer-Treat Intervention). At the county level, providers are randomized to the order/timing at which they will receive this system intervention
  Interventions: Behavioral: Screen-Refer-Treat Intervention
- Control (No Intervention): No intervention received.

INTERVENTIONS:
Behavioral: Screen-Refer-Treat Intervention — This intervention is healthcare system intervention that trains providers on validated screening tools (Online M-CHAT-R/F and STAT) and an evidence-based behavioral intervention (RIT). PCPs receive a 2-hour training workshop on the Online M-CHAT-R/F and EI Providers receive 2 day-long training workshops, one on the STAT/expedited assessment and one RIT.
  Arms: Screen-Refer-Treat Intervention

SUMMARY:
This project will implement and evaluate an innovative healthcare service delivery model designed to promote earlier access to specialized intervention for toddlers with ASD. The Screen-Refer-Treat (SRT) model provides a coordinated and cost-effective approach to early identification and intervention by involving both medical and EI providers, and represents a practical and sustainable strategy for bridging the gap between ASD concerns and ASD intervention.

DETAILED DESCRIPTION:
Although caregivers often become concerned about their child by 17-19 months of age, children do not typically receive a diagnosis of autism spectrum disorder (ASD) until they are 4½ years old, or older for Hispanic families. It is now well documented that early participation in ASD-specialized intervention can lead to significant improvements in skills and behavior for toddlers with ASD. However, despite the availability of publicly funded Part C early intervention (EI) services, long waits for a formal ASD diagnosis can prevent toddlers from receiving appropriately specialized intervention during the critical birth-to-three years. In addition, caregivers concerned about ASD experience high levels of uncertainty and stress during this waiting period. This project will implement and evaluate an innovative healthcare service delivery model designed to promote earlier access to specialized intervention for toddlers with ASD. The Screen-Refer-Treat (SRT) model provides a coordinated and cost-effective approach to early identification and intervention by involving both medical and EI providers, and represents a practical and sustainable strategy for bridging the gap between ASD concerns and ASD intervention. The SRT model, which builds on the availability of validated ASD screening tools and low-cost behaviorally-based ASD interventions, will be implemented in four diverse communities across Washington State to evaluate changes in service delivery practices for toddlers with Hispanic as well as Non-Hispanic backgrounds. The SRT model comprises three components: (1) universal ASD screening at 16-20 months and prompt referral to EI programs by primary care physicians (PCPs); (2) expedited ASD assessments within EI programs; and (3) use of an inexpensive, evidence-based ASD-specialized intervention by EI providers. An electronic version of the Modified Checklist for Autism (M-CHAT) with automated scoring that incorporates relevant follow-up questions will be provided to PCP practices, and distance coaching via telemedicine will be available to EI providers to support their ASD assessment and intervention activities. A stepped wedge cluster RCT design will be used to evaluate implementation and outcomes of the SRT model. Data on screening, referral, assessment, and intervention practices will be collected from 40 PCPs and 80 EI providers across the state prior to and following SRT implementation to identify practice changes. In addition, separate samples of caregivers of toddlers with ASD concerns (n=245) will be recruited from communities before and after SRT implementation and followed prospectively to measure differences and changes over time in caregiver wellbeing, parenting efficacy, satisfaction with healthcare systems, and toddler's social-communicative behaviors. We predict that implementation of the SRT model will be associated with higher rates of ASD screening by PCPs, earlier referral to EI programs, earlier initiation of ASD-specialized intervention, reduced time between ASD concerns and diagnosis, and improved caregiver and child outcomes.

ELIGIBILITY:
Inclusion Criteria:

PCPs:

-PCPs must work at a participating primary care practice.

EI Providers:

-EI providers must work at a participating early intervention agency.

Caregivers and Toddlers:

To be categorized as part of the ASD Concerns Sample recruited from PCP offices:

* Toddlers must demonstrate ASD risk/concern by meeting at least one of the following criteria: (1) behaviorally-based caregiver concerns about the presence of ASD; (2) behaviorally-based PCP concerns about the presence of ASD; (3) having an older sibling with an ASD diagnosis; or (4) screening positive for ASD on a validated screening tool.
* Toddlers must be between 16-20 months of age

To be categorized as part of the No ASD Concerns Sample recruited from PCP offices:

- Toddlers must be between 16-20 months of age

To be categorized as part of the ASD Dx/ASD Concerns Sample recruited from EI agencies:

* Toddlers must demonstrate ASD risk/concern by meeting at least one of the following criteria: (1) behaviorally-based caregiver concerns about the presence of ASD; (2) behaviorally-based PCP concerns about the presence of ASD; (3) having an older sibling with an ASD diagnosis; (4) screening positive for ASD on a validated screening tool; or (5) parent-report of an ASD diagnosis.
* Toddlers must be between 16-30 months of age

Exclusion Criteria:

-There are no exclusion criteria for PCPs or EI providers.

Caregivers/toddlers meeting the inclusion criteria described above will be excluded if the caregiver:

-reports that the toddler has any severe visual, auditory, or physical impairments, and/or serious medical, genetic, or neurological disorders

Min Age: 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2015-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in rates of ASD screening by PCPs at the 18-month Well-Child visit from baseline (pre-SRT intervention) to post-SRT intervention | 5 times over 4 years
  PCP self-report
Change in rates of referral for early intervention services by PCPs at the 18-month Well-Child visit from baseline (pre-SRT intervention) to post-SRT intervention | 5 times over 4 years
  PCP self-report
Change in percent of toddlers at risk for ASD recieving ASD-specialized behavioral intervention before 24 months from baseline (pre-SRT intervention) to post-SRT intervention | Every 3 months until toddlers turn 36 months of age
  Caregiver report
Change in average age at which children receive an ASD diagnosis from baseline (pre-SRT intervention) to post-SRT intervention | Every 3 months until toddlers turn 36 months of age
  Caregiver report
Change in levels of parenting stress, parenting efficacy, health quality of life, and satisfaction with the healthcare system from baseline (pre-SRT intervention) to post-SRT intervention | Every 3 months until children turn 36 months of age
  Caregiver self-report
Change in levels of pivotal social-communicative behaviors in toddlers at risk for ASD from baseline (pre-SRT intervention) to post-SRT intervention | Every 3 months until children turn 36 months of age
  Caregiver report

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Stone, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Tagavi DM, Dick CC, Attar SM, Ibanez LV, Stone WL. The implementation of the screening tool for autism in toddlers in Part C early intervention programs: An 18-month follow-up. Autism. 2023 Jan;27(1):173-187. doi: 10.1177/13623613221086329. Epub 2022 Apr 11. PMID 35403446
- [Derived] Steinman KJ, Stone WL, Ibanez LV, Attar SM. Reducing Barriers to Autism Screening in Community Primary Care: A Pragmatic Trial Using Web-Based Screening. Acad Pediatr. 2022 Mar;22(2):263-270. doi: 10.1016/j.acap.2021.04.017. Epub 2021 Apr 23. PMID 33901728
- [Derived] Ibanez LV, Stoep AV, Myers K, Zhou C, Dorsey S, Steinman KJ, Stone WL. Promoting early autism detection and intervention in underserved communities: study protocol for a pragmatic trial using a stepped-wedge design. BMC Psychiatry. 2019 Jun 7;19(1):169. doi: 10.1186/s12888-019-2150-3. PMID 31174514